CLINICAL TRIAL: NCT02257580
Title: The Effect of Intravenous E-Aminocaproic Acid (EACA) on Blood Loss and Transfusion Requirements After Bilateral Varus Rotational Osteotomy (VRO)
Brief Title: The Effect of Intravenous EACA on Blood Loss and Transfusion Requirements After Bilateral VRO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2014-303
Record Dates: First submitted 2014-09-29; First posted 2014-10-06 (Estimated); Results first posted 2022-11-23 (Actual); Last update posted 2022-11-23 (Actual); Status verified 2022-11

CONDITIONS: E-Aminocaproic Acid; Bilateral Varus Rotational Osteotomy
Keywords: E-Aminocaproic Acid; Bilateral Varus Rotational Osteotomy; Blood Loss and Transfusion; Complications; Safety
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- E-Aminocaproic acid (EACA) (Experimental): An EACA loading dose of 100 mg/kg with a max of 4-5 grams will be given up to 1 hour prior to incision. During the case, an EACA infusion of 33 mg/kg/hr (max of 1 gram/hr) will be maintained. The use of EACA will be terminated at the end of the case.
  Interventions: Drug: E-Aminocaproic acid
- Placebo (Placebo Comparator): Equivalent volume of normal saline prepared by the pharmacy.
  Interventions: Drug: E-Aminocaproic acid

INTERVENTIONS:
Drug: E-Aminocaproic acid — E-Aminocaproic acid (EACA) is a synthetic lysine analog that competitively inhibits the activation of plasminogen to plasmin and subsequently decreases the degree of fibrinolysis (Faraoni,2014} and is currently being used to decrease blood loss and transfusion requirements after orthopaedic procedures.(Eubanks,2010} Multiple meta analyses and retrospective and prospective studies have shown that EACA decreases blood loss and transfusion requirements after orthopaedic surgery{ McLeod,2013; Thompson, 2005; Thompson,2008; Gill,2008; Florentino-Pineda,2001}.Results from these studies also suggest that EACA will decreased post-operative morbidity, length of hospital stay, hospital costs, and complications.{Chimento,2013; Thompson,2005; Florentino-Pineda,2001}
  Other Names: EACA

SUMMARY:
E-Aminocaproic acid (EACA) is an anti-fibrinolytic agent that is used to decrease blood loss and transfusion requirements after several orthopedic procedures. The aim of this prospective double-blind placebo-controlled randomized trial is to determine whether IV EACA reduces intra-operative calculated total blood loss in patients undergoing bilateral varus rotational osteotomy (VRO). This study will also investigate intraoperative cell saver utilization, transfusion of allogeneic blood, hospital length-of-stay (LOS), short term complications, and long-term outcomes.This study will provide Level I evidence and has the potential to improve outcomes in children undergoing this procedure.

DETAILED DESCRIPTION:
The participating anesthesiologists will not be blinded to study arms and hypotheses. Dr. Christopher Edmonds will be the head anesthesiologist for this study and will administer anesthetics to participants in this trial whenever his schedule makes it possible. Anesthesia will be conducted in a standardized fashion, with IV sedation using Versed and IV propofol, +/- Fentanyl and Ketamine . A Combined Spinal-Epidural (CSE) will be placed using 12.5-20 mg of bupivacaine. If a CSE is unsuccessful and an epidural and/or spinal are successfully obtained, the patient may still be included in the study. Patients not receiving neuraxial anesthesia will be excluded. If a patient requires general anesthesia, it will be induced at this time, but the patient will be excluded from the study. An arterial line and additional venous access will be obtained in standardized sterile practice. Sedation will be maintained with IV propofol. IV Valium, Toradol and IV acetaminophen will be given towards the end of the case, per anesthesiologist's discretion.

The blood pressure target will be 20-25% below baseline, which will be achieved primarily with the neuraxial anesthesia. For blood pressure above this range, the epidural will be dosed with a short-acting local anesthetic, and/or IV sedation will be titrated as per the anesthesiologist's judgment. For hypotension below this range, pressors or intravenous pressors will be given. An IV fluid bolus may also be given in the amount of 10-20cc/kg. Additional maintenance IV fluids will be given to maintain urine output of at least 0.5-1ml/kg/hr. The criteria for transfusion of blood products will be a hemoglobin level of < 7.0 g/dL or a hemoglobin level of < 10.0 g/dL with clinical signs of symptomatic anemia (e.g., unexplained tachycardia, hypotension unresponsive to fluids or vasopressors, change in mental status, low urine output, and shortness of breath). Blood will be administered 1 unit at a time, and the presence of symptoms or signs will be reassessed after each unit. This algorithm may be altered by the treating physician (e.g., PACU attending, surgeon, or the OR anesthesiologist), however all decisions will be supported by reasonable documentation. Drains will be removed on POD 2 unless specified by the attending surgeon. Of note, the chart of the patient will clearly indicate him/her as a study patient; a sticker will be place on the front of each participating patient's chart. Their enrollment will also be communicated in the clinician rounding notes for each patient. Drains will be labeled for each study participant as well, and nurses will record the drain outputs per their floor protocol.

Attending surgeons, orthopedic surgery residents, physician assistants and research assistants involved with this study will assist in data collection. For each patient, we will collect demographic data, pre-operative CBC data, intra-operative cell saver auto-transfusion volumes, post-operative number of packed red blood cell units transfused, post-operative CBC data, post-operative drain outputs, and post-operative complications. This information will be gathered from the peri-operative medical records and electronic medical records. Surgeons and clinical and research personnel will review medical chart and progress notes for evidence of clinically significant VTE, reoperation, hematoma, seroma, and infection.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for bilateral varus rotational osteotomy (VRO) with or without associated soft tissue and osseous procedures

Exclusion Criteria:

* Preoperative use of an anticoagulant (Plavix, warfarin, lovenox, etc.)
* History of hypersensitivity to EACA
* History of thromboembolic event (e.g., PE or DVT)
* History of renal insufficiency or failure
* Congenital or acquired coagulopathy as evidence by INR >1.4 or PTT > 1.4 times normal, or Platelets <150,000/mm3 on preoperative laboratory testing
* Use of hormone replacement therapy or hormonal contraceptive agents within days prior to surgery
* Use of acetylsalicylic acid (ASA), antiplatelet agents within 7 days prior to surgery
* Pregnant
* Breastfeeding
* Not received neuraxial anesthesia

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 28 (Actual)
Dates: Start 2015-04-01 (Actual); Primary Completion 2020-10-26 (Actual); Study Completion 2020-10-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Scher, MD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Eubanks JD. Antifibrinolytics in major orthopaedic surgery. J Am Acad Orthop Surg. 2010 Mar;18(3):132-8. PMID 20190103
- [Background] Faraoni D, Goobie SM. The efficacy of antifibrinolytic drugs in children undergoing noncardiac surgery: a systematic review of the literature. Anesth Analg. 2014 Mar;118(3):628-36. doi: 10.1213/ANE.0000000000000080. PMID 24557107
- [Background] McLeod LM, French B, Flynn JM, Dormans JP, Keren R. Antifibrinolytic Use and Blood Transfusions in Pediatric Scoliosis Surgeries Performed at US Children's Hospitals. J Spinal Disord Tech. 2015 Oct;28(8):E460-6. doi: 10.1097/BSD.0b013e3182a22a54. PMID 24091932
- [Background] Thompson GH, Florentino-Pineda I, Poe-Kochert C. The role of amicar in decreasing perioperative blood loss in idiopathic scoliosis. Spine (Phila Pa 1976). 2005 Sep 1;30(17 Suppl):S94-9. doi: 10.1097/01.brs.0000175188.05542.a9. PMID 16138073
- [Background] Thompson GH, Florentino-Pineda I, Poe-Kochert C, Armstrong DG, Son-Hing J. Role of Amicar in surgery for neuromuscular scoliosis. Spine (Phila Pa 1976). 2008 Nov 15;33(24):2623-9. doi: 10.1097/BRS.0b013e318187c046. PMID 18981961
- [Background] Gill JB, Chin Y, Levin A, Feng D. The use of antifibrinolytic agents in spine surgery. A meta-analysis. J Bone Joint Surg Am. 2008 Nov;90(11):2399-407. doi: 10.2106/JBJS.G.01179. PMID 18978408
- [Background] Florentino-Pineda I, Blakemore LC, Thompson GH, Poe-Kochert C, Adler P, Tripi P. The Effect of epsilon-aminocaproic acid on perioperative blood loss in patients with idiopathic scoliosis undergoing posterior spinal fusion: a preliminary prospective study. Spine (Phila Pa 1976). 2001 May 15;26(10):1147-51. doi: 10.1097/00007632-200105150-00011. PMID 11413428
- [Background] Chimento GF, Huff T, Ochsner JL Jr, Meyer M, Brandner L, Babin S. An evaluation of the use of topical tranexamic acid in total knee arthroplasty. J Arthroplasty. 2013 Sep;28(8 Suppl):74-7. doi: 10.1016/j.arth.2013.06.037. PMID 24034510

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients aged 18 or younger with CP indicated for bilateral VRO. Hx of a thromboembolic event, renal insufficiency or failure, known hypersensitivity to EACA, congenital or acquired coagulopathy, pts that could not receive neuraxial anesthesia, being treated with anticoagulants, hormone replacement therapy or hormonal contraceptive agent were excluded. Pts undergoing bilateral VRO were identified and screened by the study surgeons. 2 screened pts declined to participate, 2 did not qualify.
Period: Overall Study
Arm/Group | E-Aminocaproic Acid (EACA) | Placebo
Started | 16 | 12
Completed | 16 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | E-Aminocaproic Acid (EACA) | Placebo | Total
Number analyzed (Participants) | 16 | 12 | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 16 | 12 | 28
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 10
  Male | 10 | 8 | 18
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 16 | 12 | 28

OUTCOME MEASURES:

1. Primary Outcome: Intraoperative Calculated Total Blood Loss
Description: Determined by estimated blood volume, calculated using difference in preoperative and postoperative hemoglobin and applied to the Nadler equation for estimating blood volume while adjusting for transfused hemoglobin to produce a single metric of calculated intraoperative blood loss.
Time Frame: Intraoperative (3-6 hours)
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | E-Aminocaproic Acid (EACA) | Placebo
Number analyzed (Participants) | 16 | 12
mL | 535.7 (356.6) | 628.0 (235.8)

2. Secondary Outcome: Intraoperative Cell Saver Utilization
Description: Number of participants requiring 1 unit of intraoperative cell saver transfusion. Patients either received or did not receive intraoperative cell saver transfusion. The maximum number of intraoperative units transfused in this study was 1 unit. The count of participants in the data table refers to the number of patients who received this transfusion.
Time Frame: Intraoperative, 1 day
Measure: Count of Participants; unit: Participants
Arm/Group | E-Aminocaproic Acid (EACA) | Placebo
Number analyzed (Participants) | 16 | 12
Participants | 7 | 7

3. Secondary Outcome: Postoperative Allogeneic Blood Transfusion
Description: The number of participants that required 1 unit of blood transfused post-operatively. Patients received blood if necessary post operatively, and the maximum number of units a patient received was 1. The count of participants refers to the number of patients who received this transfusion unit.
Time Frame: Post-Surgery, an expected average of 1 week
Measure: Count of Participants; unit: Participants
Arm/Group | E-Aminocaproic Acid (EACA) | Placebo
Number analyzed (Participants) | 16 | 12
Participants | 4 | 3

4. Secondary Outcome: Post Operative Blood Loss
Description: 24 hour drain output (mL)
Time Frame: Post-Surgery, 24 hours
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | E-Aminocaproic Acid (EACA) | Placebo
Number analyzed (Participants) | 16 | 12
mL | 72.5 (69.8) | 103.3 (91.4)

5. Secondary Outcome: Length of Hospital Stay
Description: postoperative day of discharge after surgery- day of intake.
Time Frame: Post-Surgery, an expected average of 1 week
Measure: Mean (Full Range); unit: days
Arm/Group | E-Aminocaproic Acid (EACA) | Placebo
Number analyzed (Participants) | 16 | 12
days | 5.5 [4 to 7] | 5.1 [4 to 6]

6. Secondary Outcome: Complications [VTE (Symptomatic of DVT or PE), Infection (Superficial, Deep), Hematoma, Seroma, Reoperation, and Death]
Description: Incidence of VTE (symptomatic of DVT or PE), infection (superficial, deep), hematoma, seroma, reoperation, and death, measured in person-years ( x cases per 100,000 person years)
Time Frame: an expected average of 1 week (post-surgery), Follow-up at 6 weeks
Measure: Number; unit: cases per 100,000 person years
Arm/Group | E-Aminocaproic Acid (EACA) | Placebo
Number analyzed (Participants) | 16 | 12
cases per 100,000 person years | 0 | 0

ADVERSE EVENTS:
Time Frame: Day of surgery through 6 weeks post-op.
Arm/Group | E-Aminocaproic Acid (EACA) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/12
Other Adverse Events (participants affected / at risk) | 0/16 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2014-12-10): https://cdn.clinicaltrials.gov/large-docs/80/NCT02257580/Prot_SAP_000.pdf
  • Informed Consent Form (2014-12-09): https://cdn.clinicaltrials.gov/large-docs/80/NCT02257580/ICF_001.pdf